CLINICAL TRIAL: NCT05364528
Title: Pregnancy Rate in Single Step Versus After Load Technique of Embryo Transfer: a Retrospective Analysis
Brief Title: Pregnancy Rate in Direct Versus Afterload Technique of Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 12022
Record Dates: First submitted 2022-05-03; First posted 2022-05-06 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Fertility Issues; IVF; Embryo Transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clinical pregnancies with direct catheter: Clinical pregnancies occurred after fresh and frozen blastocyst transfers using direct technique.
- clinical pregnancies with afterload catheter: Clinical pregnancies occurred after fresh and frozen blastocyst transfers using afterload technique.

SUMMARY:
The primary outcome of the study is to determine if a difference in terms of pregnancy rate exists between direct and afterload embryo transfer (ET) techniques.

The secondary end points include the evaluation of the difficult transfer rates.

DETAILED DESCRIPTION:
The study database includes all the single fresh and frozen (G5-G6) blastocyst transfers performed at Humanitas Fertility Centre between 1st January 2016 and 31th December 2021 by using the direct and afterload protocols.

Any blastocysts that underwent preimplantation genetic testing will be excluded from the analysis, as well as embryos derived from gamete donation or those imported from other centers.

Data are gathered using a specific internal web-based database, which allows to organize, store and readily retrieve information about patients and IVF cycle.

ELIGIBILITY:
Inclusion Criteria:

* IVF procedure
* Fresh and frozen single blastocyst transfer

Exclusion Criteria:

* Any blastocysts that underwent PGS testing
* Embryos derived from gamete donation
* Embryos imported from other centers

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study database includes all the single fresh and frozen (G5-G6) blastocyst transfers performed at Humanitas Fertility Centre between 1st January 2016 and 31th December 2021 by using the direct and afterload protocols.
Sampling Method: Non-Probability Sample
Enrollment: 8127 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 6 years
  number of pregnancies diagnosed by ultrasonographic visualization of one or more gestational sacs x 100 divided by the number of embryo transfer cycles

SECONDARY OUTCOMES:
difficult transfer rate | 6 years
  advancement of the outer sheath, multiple attempts, force, required manipulation, use of a stylet or tenaculum, dilatation, use of a different catheter

REFERENCES:
- [Derived] Cirillo F, Immediata V, Ronchetti C, Carletti T, Morenghi E, Albani E, Baggiani A, Levi-Setti PE. Steps forward in embryo transfer technique: a retrospective study comparing direct versus afterload catheters at different time frames. J Assist Reprod Genet. 2023 Dec;40(12):2895-2902. doi: 10.1007/s10815-023-02957-y. Epub 2023 Oct 11. PMID 37819552